CLINICAL TRIAL: NCT02859116
Title: Collection of Gastrointestinal Tissue Samples for the Characterization and ex Vivo Functional Assessment of Chemoreceptors
Acronym: ISTAR-T
Status: Completed | Type: Observational
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: TRIMD FH 794609
Record Dates: First submitted 2016-07-13; First posted 2016-08-08 (Estimated); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Diabetes
Keywords: Metabolic diseases
MeSH Terms: conditions — Diabetes Mellitus; Metabolic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of tissues from the digestive system of patients undergoing surgery for clinical purposes. Tissue samples will be used to assess a mechanism of action (MOA) for the regulation of gut hormone secretion and nutrient absorption. Patients will be also asked to provide clinical/medical data and blood samples prior to their surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Collection of digestive tissues: Digestive tissues will be collected from participants undergoing scheduled (non-emergent) gastrointestinal surgery.
  Interventions: Procedure: Collection of digestive tissues

INTERVENTIONS:
Procedure: Collection of digestive tissues — The surgeon will resect a sample (approximately 1-5 cm x 1-5 cm) of healthy tissue from the distal margins of the segment and at least 4 cm from the diseased area. The specimen for research will be obtained from the tissue that would ordinarily be removed during surgery.The tissue collected for our research purposes will be only remnant tissue which is discarded by the surgeon during the surgical intervention and has no diagnostic clinical value.

SUMMARY:
The purpose of this study is to help scientists understand how the gut senses ingested nutrients and what kind of processes take place for their absorption in order to establish the association with diabetes and other metabolic diseases Scientists need human specimens to study.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 18 years and older who are having elective gastrointestinal surgery
2. Able to provide written, informed consent

Exclusion Criteria:

1. Unable to provide written, informed consent
2. Use of antibiotics for more than 5 consecutive days in the three months prior to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective gastrointestinal surgical procedures by the surgeons of the Center for Specialized Surgery.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2016-07-21 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Tissue collection | Day of surgery
  During surgery, a tissue specimen that would normally be discarded, will be obtained and used to identify the localization and amount of different proteins that regulate nutrient absorption.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Pratley, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adler E, Hoon MA, Mueller KL, Chandrashekar J, Ryba NJ, Zuker CS. A novel family of mammalian taste receptors. Cell. 2000 Mar 17;100(6):693-702. doi: 10.1016/s0092-8674(00)80705-9. PMID 10761934
- [Background] Chandrashekar J, Hoon MA, Ryba NJ, Zuker CS. The receptors and cells for mammalian taste. Nature. 2006 Nov 16;444(7117):288-94. doi: 10.1038/nature05401. PMID 17108952
- [Background] Chandrashekar J, Mueller KL, Hoon MA, Adler E, Feng L, Guo W, Zuker CS, Ryba NJ. T2Rs function as bitter taste receptors. Cell. 2000 Mar 17;100(6):703-11. doi: 10.1016/s0092-8674(00)80706-0. PMID 10761935
- [Background] Margolskee RF, Dyer J, Kokrashvili Z, Salmon KS, Ilegems E, Daly K, Maillet EL, Ninomiya Y, Mosinger B, Shirazi-Beechey SP. T1R3 and gustducin in gut sense sugars to regulate expression of Na+-glucose cotransporter 1. Proc Natl Acad Sci U S A. 2007 Sep 18;104(38):15075-80. doi: 10.1073/pnas.0706678104. Epub 2007 Aug 27. PMID 17724332
- [Background] Wu SV, Rozengurt N, Yang M, Young SH, Sinnett-Smith J, Rozengurt E. Expression of bitter taste receptors of the T2R family in the gastrointestinal tract and enteroendocrine STC-1 cells. Proc Natl Acad Sci U S A. 2002 Feb 19;99(4):2392-7. doi: 10.1073/pnas.042617699. PMID 11854532
- [Background] Deshpande DA, Wang WC, McIlmoyle EL, Robinett KS, Schillinger RM, An SS, Sham JS, Liggett SB. Bitter taste receptors on airway smooth muscle bronchodilate by localized calcium signaling and reverse obstruction. Nat Med. 2010 Nov;16(11):1299-304. doi: 10.1038/nm.2237. Epub 2010 Oct 24. PMID 20972434
- [Background] Kinnamon SC. Taste receptor signalling - from tongues to lungs. Acta Physiol (Oxf). 2012 Feb;204(2):158-68. doi: 10.1111/j.1748-1716.2011.02308.x. Epub 2011 May 7. PMID 21481196
- [Background] Jang HJ, Kokrashvili Z, Theodorakis MJ, Carlson OD, Kim BJ, Zhou J, Kim HH, Xu X, Chan SL, Juhaszova M, Bernier M, Mosinger B, Margolskee RF, Egan JM. Gut-expressed gustducin and taste receptors regulate secretion of glucagon-like peptide-1. Proc Natl Acad Sci U S A. 2007 Sep 18;104(38):15069-74. doi: 10.1073/pnas.0706890104. Epub 2007 Aug 27. PMID 17724330
- [Background] Steinert RE, Gerspach AC, Gutmann H, Asarian L, Drewe J, Beglinger C. The functional involvement of gut-expressed sweet taste receptors in glucose-stimulated secretion of glucagon-like peptide-1 (GLP-1) and peptide YY (PYY). Clin Nutr. 2011 Aug;30(4):524-32. doi: 10.1016/j.clnu.2011.01.007. Epub 2011 Feb 15. PMID 21324568
- [Background] Jeon TI, Zhu B, Larson JL, Osborne TF. SREBP-2 regulates gut peptide secretion through intestinal bitter taste receptor signaling in mice. J Clin Invest. 2008 Nov;118(11):3693-700. doi: 10.1172/JCI36461. Epub 2008 Oct 9. PMID 18846256
- [Background] Chandra R, Liddle RA. Cholecystokinin. Curr Opin Endocrinol Diabetes Obes. 2007 Feb;14(1):63-7. doi: 10.1097/MED.0b013e3280122850. PMID 17940422
- [Background] Chao CY, Huang CJ. Bitter gourd (Momordica charantia) extract activates peroxisome proliferator-activated receptors and upregulates the expression of the acyl CoA oxidase gene in H4IIEC3 hepatoma cells. J Biomed Sci. 2003 Nov-Dec;10(6 Pt 2):782-91. doi: 10.1159/000073966. PMID 14631118
- [Background] Kim KS, Egan JM, Jang HJ. Denatonium induces secretion of glucagon-like peptide-1 through activation of bitter taste receptor pathways. Diabetologia. 2014 Oct;57(10):2117-25. doi: 10.1007/s00125-014-3326-5. Epub 2014 Jul 13. PMID 25016595
- [Background] Kyriazis GA, Smith KR, Tyrberg B, Hussain T, Pratley RE. Sweet taste receptors regulate basal insulin secretion and contribute to compensatory insulin hypersecretion during the development of diabetes in male mice. Endocrinology. 2014 Jun;155(6):2112-21. doi: 10.1210/en.2013-2015. Epub 2014 Apr 8. PMID 24712876
- [Background] Kyriazis GA, Soundarapandian MM, Tyrberg B. Sweet taste receptor signaling in beta cells mediates fructose-induced potentiation of glucose-stimulated insulin secretion. Proc Natl Acad Sci U S A. 2012 Feb 21;109(8):E524-32. doi: 10.1073/pnas.1115183109. Epub 2012 Feb 6. PMID 22315413
- [Background] Nakagawa Y, Nagasawa M, Yamada S, Hara A, Mogami H, Nikolaev VO, Lohse MJ, Shigemura N, Ninomiya Y, Kojima I. Sweet taste receptor expressed in pancreatic beta-cells activates the calcium and cyclic AMP signaling systems and stimulates insulin secretion. PLoS One. 2009;4(4):e5106. doi: 10.1371/journal.pone.0005106. Epub 2009 Apr 8. PMID 19352508
- [Background] Drewnowski A, Gomez-Carneros C. Bitter taste, phytonutrients, and the consumer: a review. Am J Clin Nutr. 2000 Dec;72(6):1424-35. doi: 10.1093/ajcn/72.6.1424. PMID 11101467
- [Background] Bachmanov AA, Beauchamp GK. Taste receptor genes. Annu Rev Nutr. 2007;27:389-414. doi: 10.1146/annurev.nutr.26.061505.111329. PMID 17444812
- See also: Translational Research Institute for Metabolism and Diabetes — http://www.tri-md.org/